CLINICAL TRIAL: NCT00652119
Title: Pilot Trial of Intraperitoneal Paclitaxel and Carboplatin With IV Avastin Therapy in Treatment of Women With Newly Diagnosed, Optimally Cytoreduced Carcinoma of Mullerian Origin
Brief Title: Intraperitoneal Paclitaxel and Carboplatin With IV Avastin Therapy in Patients With Carcinomas of Mullerian Origin
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Genentech, Inc. (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Richard Thomas Penson, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-426; NCI-2010-00091 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2008-03-31; First posted 2008-04-03 (Estimated); Last update posted 2020-08-19 (Actual); Status verified 2020-08

CONDITIONS: Ovarian Cancer; Peritoneal Cancer; Fallopian Tube Cancer
Keywords: Ovarian Cancer; Peritoneal Cancer; Fallopian Tube Cancer; Carcinoma of Mullerian Origin; Paclitaxel; Taxol; Carboplatin; Paraplatin®; Avastin; Bevacizumab; Anti-VEGF monoclonal antibody; rhuMAb-VEGF
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — Paclitaxel; Carboplatin; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Paclitaxel + Carboplatin + Avastin (Experimental): Paclitaxel Cycle 1 = 60 mg/m^2 IV weekly over 1 hour x 3 weeks; Cycles 2-6 = 60 mg/m^2 IP weekly over 1 hour x 3 weeks of each cycle.
  Carboplatin Cycle 1 = AUC 6 IV over 1 hour on day 1; Cycles 2-6 = AUC 6 IP over 1 hour on day 1 of each cycle.
  Avastin Cycle 2 = 15 mg/kg IV over 90 minutes on day 8; Cycles 3-6 = 15 mg/kg IV on day 1 of each cycle.
  Interventions: Drug: Paclitaxel; Drug: Carboplatin; Drug: Avastin

INTERVENTIONS:
Drug: Paclitaxel — Cycle 1 = 60 mg/m^2 IV weekly over 1 hour x 3 weeks; Cycles 2-6 = 60 mg/m^2 IP weekly over 1 hour x 3 weeks of each cycle.
  Other Names: Taxol
Drug: Carboplatin — Cycle 1 = AUC 6 IV over 1 hour on day 1; Cycles 2-6 = AUC 6 IP over 1 hour on day 1 of each cycle.
  Other Names: Paraplatin®
Drug: Avastin — Cycle 2 = 15 mg/kg IV over 90 minutes on day 8; Cycles 3-6 = 15 mg/kg IV on day 1 of each cycle.
  Other Names: Bevacizumab; Anti-VEGF monoclonal antibody; rhuMAb-VEGF

SUMMARY:
The goal of this clinical research study is to learn about the safety and tolerability of paclitaxel and carboplatin when given in combination with Avastin to patients with ovarian, primary peritoneal, or fallopian tube cancer.

Objectives:

Primary study goals:

To investigate the safety and tolerability of carboplatin and paclitaxel administered IP in combination with IV Avastin To determine if Avastin influences the pharmacokinetics of IP administered chemotherapeutic agents

Secondary study goals:

To determine the systemic exposure to paclitaxel and carboplatin during initial and late cycles of IP dosing.

To collect overall survival (OS) and progression-free survival (PFS) To determine changes in IP VEGF levels To determine site of first recurrence Information on CA-125 response and clinical response will be descriptive as secondary goals of this study

Exploratory goal:

To estimate proportion of patients completing entire course of treatment

DETAILED DESCRIPTION:
The Study Drugs:

Carboplatin is designed to interfere with the growth of cancer cells by stopping cell division, which may cause the cells to die.

Paclitaxel is designed to block the mechanisms of cell division in cancer cells, which may cause them to die.

Avastin is designed to prevent or slow down the growth of cancer cells by blocking the effects of VEGF, a blood-vessel stimulating agent that plays an important role in the growth of both normal and abnormal blood vessels.

Intraperitoneal Port (IP) Placement:

If you are found eligible to take part in this study, you will need to have an IP port, called an intraperitoneal catheter tube, placed into the abdomen. The catheter will be used to give the paclitaxel and carboplatin directly into your abdomen. You may already have had this catheter placed at a previous surgery. If not, you will have a minor surgical procedure in the operating room to have it placed. You will be asked to sign a separate surgical consent form describing this procedure, the risks involved, and the steps for taking care of the catheter while it is in place.

Study Drug Administration:

You will receive up to 6 cycles of treatment with the study drugs. Each cycle is 21 days (3 weeks) long.

Cycle 1:

You will receive paclitaxel and carboplatin through a needle in your vein on Day 1. Paclitaxel is given first followed by carboplatin. Both drugs are given over 1 hour. On Days 8 and 15 you will only receive paclitaxel by vein. This infusion is also given over 1 hour.

Cycle 2:

On Day 1, about 2 cups of normal saline will be infused into your abdomen through the IP catheter. This infusion takes 30-60 minutes. You will then receive paclitaxel through the IP port in your abdomen. When the paclitaxel infusion is complete, you will receive carboplatin through the IP port. Each infusion takes about 1 hour. After the chemotherapy infusions are complete, another 2-4 cups of normal saline will be infused through the port. This is done to help move the chemotherapy to all areas of your abdomen. You will be asked to change position frequently.

On Day 8, about 2 cups of normal saline will be infused into your abdomen through the IP catheter. You will then receive paclitaxel through the IP port in your abdomen over 1 hour. While you are receiving paclitaxel through your IP port, you will also receive Avastin by vein. The first dose of Avastin will be given over 90 minutes. If you tolerate the first infusion well, the second infusion (given in Cycle 3) may be given over 60 minutes. If the 60-minute infusion is well-tolerated, all infusions after that may be given over 30 minutes. After the paclitaxel infusion is complete, you will receive another 2-4 cups of normal saline through the port. You will be asked to change position frequently.

On Day 15, about 2 cups of normal saline will be infused into your abdomen through the IP catheter. You will then receive paclitaxel through the IP port in your abdomen. After the paclitaxel infusion is complete, you will receive another 2-4 cups of normal saline through the port. You will be asked to change position frequently.

Cycles 3-6:

On Day 1, about 2 cups of normal saline will be infused into your abdomen through the IP catheter. You will receive paclitaxel through the IP catheter over 1 hour. After completing paclitaxel, you will receive carboplatin through the IP catheter over 1 hour. After these infusions are complete you will receive another 2-4 cups of normal saline through the port. You will be asked to change position frequently. While undergoing IP therapy with paclitaxel and carboplatin, you will also receive the second infusion of Avastin by vein. The length of this infusion will depend how well you tolerated the drug the first time it was given in Cycle 2.

On Days 8 and 15, about 2 cups of normal saline will be infused into your abdomen through the IP catheter. You will then receive paclitaxel through the IP port in your abdomen over 1 hour. After the paclitaxel infusion is complete, you will receive another 2-4 cups of normal saline through the port. You will be asked to change position frequently.

Before you receive paclitaxel and carboplatin, you will receive the drug dexamethasone by vein to help decrease the risk of study drug side effects. You may also receive other drugs (such as cimetidine and diphenhydramine) by vein to help with side effects, such as nausea and allergic reaction. The choice of which drugs to use is up to your doctor.

Study Visits:

On Day 1 of each cycle, the following tests and procedures will be performed:

* Your medical history will be recorded, including a list of any drugs you are taking.
* You will be asked how well you are able to perform your normal daily activities (performance status evaluation).
* You will have physical exam, measurement of your vital signs, and a neurological exam.
* You will be asked about any side effects you are experiencing.
* Blood (about 3 teaspoons) will be drawn for routine tests (this will be repeated on Days 8 and 15 of each cycle as well).

Blood (about 1 teaspoon) will be drawn to check your CA125 level before treatment starts in Cycle 1 and on Day 1 of Cycles 2, 4, and 6.

Before treatment starts in Cycle 1 and on Day 8 of Cycle 2 and Day 1 of Cycles 3-6, urine will be collected for routine tests.

On Days 1, 8, and 15 of Cycles 1, 2, and 4, blood (1 teaspoon each time) will be drawn 12 different times each day for pharmacokinetic (PK) testing. PK testing measures the amount of study drugs in the body at different time points. Blood (1 teaspoon each time) will also be drawn 1 time on Days 2 and 3 of Cycles 1, 2, and 4.

On Day 8 of Cycle 2 and Day 1 of Cycles 3, 4, and 6 before paclitaxel starts, you will have the levels of vascular endothelial growth factor (VEGF) in your abdominal fluid measured. VEGF is a protein that causes fluid build-up (ascites) in the abdomen. About 2 cups of normal saline will be infused through the IP port. You will be asked to change positions for about 15 minutes. Then about 3-4 tablespoons of the fluid will be removed from the port with a syringe. This shows how Avastin is affecting your abdominal fluid. You will also have blood (about 1 teaspoon) drawn to check the levels of VEGF in your blood.

Length of Study:

You may remain on this study for up to 6 cycles. You will be taken off study early if the disease gets worse or intolerable side effects occur.

End-of-Study Visit:

Once you are off study, you will have an end-of-study visit. At this visit, the following tests and procedures will be performed:

* You will have a physical exam.
* You will have a computed tomography (CT) scan.
* Blood (about 1 teaspoon) will be drawn to check your CA125 level.

Long-Term Follow-Up:

After your last study visit, you will be contacted about every 3 months from then on to check on how you are doing. You will return to the clinic or researchers will call you on the phone to ask you questions about how you are doing. Your doctor will tell you if any standard tests and procedures need to be performed.

This is an investigational study. Avastin, carboplatin, and paclitaxel are FDA approved and commercially available for the treatment of many types of cancer. At this time, the addition of Avastin to paclitaxel and carboplatin is being used to treat ovarian cancer in research only.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed epithelial carcinoma of mullerian origin. Specifically, ovarian, primary peritoneal and tubal carcinoma will be allowed. All histologic subtypes are eligible.
2. Stage III or IV disease. Stage IV disease by virtue of pleural effusions is allowed but stage IV disease with visceral metastases e.g. lung, liver or abdominal wall is NOT ELIGIBLE. Please discuss any eligibility concerns directly with the P.I., Dr. Richard Penson.
3. Patient must have undergone surgical staging and debulking with optimal (less than 1cm) cytoreduction.
4. No significant intra-abdominal adhesions or other contraindication to IP port placement.
5. Patients must give written informed consent.
6. Patient must be age 18 years or older.
7. Adequate bone marrow function with an ANC greater that 2,500 and Platelets greater than 100,000 cubic millimeters.
8. No proteinuria or less than +1; if greater, 24-hour urine collection must be performed to document less than or equal to 1gm/24 hours of protein.
9. ECOG performance status less than or equal to 1.

Exclusion Criteria:

1. Visible disease on post-operative imaging (recognizing the limitations of postoperative CT scans due to postoperative changes there should be unequivocal CT evidence of residual disease greater than 1cm)
2. ECOG performance status greater than or equal to 2
3. Previous chemotherapy for the disease under study
4. Suboptimal (greater than 1 cm residual disease) cytoreduction
5. Creatinine greater than 1.5 mg/dL
6. SGOT greater than 2 x ULN, bilirubin greater than 1.5 x ULN
7. Colostomy or ileostomy
8. Concurrent invasive malignancy. (Patients with concurrent superficial endometrial carcinoma are eligible if their endometrial carcinoma is superficial or invades less than 50% the thickness of the myometrium.)
9. Known hypersensitivity to E.coli derived products or to any component of Avastin
10. Active psychiatric or mental illness that makes informed consent or careful clinical follow-up unlikely
11. History of myocardial infarction within 6 months
12. History of stroke or transient ischemia attack within 6 months
13. Inadequately controlled hypertension greater than 140/90 mm Hg on antihypertensive medication(s)
14. Any prior history of hypertensive crisis or hypertensive encephalopathy
15. Clinically significant peripheral vascular disease
16. Significant vascular disease (e.g. aortic aneurysm, aortic dissection)
17. Unstable angina
18. New York Heart Association (NYHA) grade II or greater congestive heart failure
19. Evidence of coagulopathy or bleeding diathesis
20. Known central nervous system disease or brain metastases
21. Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to day 28 (first dose of Avastin), anticipation of need for major surgical procedure during the course of the study
22. Minor surgical procedures such as fine needle aspirations or core biopsies or laparoscopy for IP catheter placement within 7 days prior to cycle 2 day 8
23. Open wound, ulcer, or bone fracture
24. History of abdominal fistula, gastrointestinal perforation or intra-abdominal abscess; current signs and symptoms of bowel obstruction; current dependency on IV hydration or TPN
25. Pregnant (positive pregnancy test) or lactating

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2008-02 (Actual); Primary Completion 2009-08 (Actual); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Number of Patients Who Complete Entire Treatment Course | Total treatment course = 6 cycles (1 cycle is 21 days)
  Rate of completers estimated along with a 95% confidence interval to evaluate the tolerability of this regimen.
Systemic Exposure to Paclitaxel and Carboplatin | Second and fourth 21 day cycle
  Primary objective of pharmacokinetic studies is to determine whether rate and extent absorption of paclitaxel and carboplatin into systemic circulation when given by the intraperitoneal port (IP) route is influenced by concurrent administration of Avastin by vein. Sampling to define plasma concentration time courses of paclitaxel and carboplatin performed during second cycle without Avastin and fourth cycle of therapy with Avastin. Pharmacokinetic parameters and variables calculated according to standard equations. Concentration-time profiles of carboplatin and its metabolites analyzed by noncompartmental methods and/or nonlinear least squares regression. Mean values of pharmacokinetic parameters statistically compared using the two-tailed t-test.

SECONDARY OUTCOMES:
Median Progression Free Survival | From the start of treatment until the time of death or progression, up to 10 years
Median Overall Survival | From the start of treatment until the time of death, up to 20 years
Change in Intraperitoneal VEGF levels | Cycle 4-6 day 8, day 1 of cycles 7-12 and 16-18 (cycle is 21 days)
Site of Cancer First Recurrence | At the time of first recurrence, assessed up to 10 years
Change in Plasma CA-125 Level | 1 Year
Clinical Response Rate | 1 Year
  The number of participants that achieved a clinical response following treatment. Clinical response is defined as achieving a best overall response of a complete response (CR) or a partial response (PR).
  * Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
  * Partial Response (PR): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.

CONTACTS AND LOCATIONS:
Overall Officials: Richard T Penson, MD, Principal Investigator — Massachusetts General Hospital
Locations (5):
- United States (5):
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Fred Hutchinson Cancer Research Center, Seattle, Washington